CLINICAL TRIAL: NCT02526771
Title: A Randomized Controlled Study of Conventional or Unconventional Lymph Node Dissection During Resection of Intrahepatic Cholangiocarcinoma
Brief Title: Conventional or Unconventional Lymph Node Dissection During Resection of Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHLND-2015-8-10
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: lymph node dissection
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional lymph node dissection (Experimental): conventional lymph node dissection during resection of intrahepatic cholangiocarcinoma
  Interventions: Procedure: conventional lymph node dissection
- unconventional lymph node dissection (Active Comparator): unconventional lymph node dissection during resection of intrahepatic cholangiocarcinoma
  Interventions: Procedure: unconventional lymph node dissection

INTERVENTIONS:
Procedure: conventional lymph node dissection — conventional lymph node dissection during resection of intrahepatic cholangiocarcinoma
  Arms: conventional lymph node dissection
Procedure: unconventional lymph node dissection — unconventional lymph node dissection during resection of intrahepatic cholangiocarcinoma
  Arms: unconventional lymph node dissection

SUMMARY:
The aim of this study is to compare the surgical outcomes of conventional lymph node dissection with unconventional lymph node dissection during resection of Intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) is one of the primary liver cancer, which has higher malignant, more difficult treatment and worse prognosis compared to hepatocellular carcinoma and its incidence continues to rise. The main radical treatment is surgical resection, however, postoperative recurrence rate is extremely high. The 3-year recurrence rate is more than 50%. It is reported that lymph node metastasis rate of ICC is as high as 20% to 65%, which is the most significant factor of the poor prognosis. The probability of lymph node metastasis is 13% when lymph nodes metastasis were not found preoperative or intraoperative. It is highly controversial whether or not to undergo conventional lymph node dissection when lymph nodes metastasis were not found preoperative or intraoperative . A number of researchers approved of lymph node dissection at that situation. However, some authors such as Kim suggest that lymph node resection is not necessary. Others such as Yang think should consider in different condition. Clark CJ thinks that the evidence for dissection or not of lymph node is insufficient in view of the above reasons, the investigators have planned to implement a randomized controlled study to confirm the prognostic value of conventional or unconventional lymph node dissection during resection of Intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* Diagnosis of intrahepatic cholangiocarcinoma ( through imaging, serology, intraoperative frozen, etc.)
* No lymph node metastasis preoperatively or intraoperatively.
* Tumors can be completely resected.
* Criteria of liver function: Child A-B level, serum bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
* Patients who can understand this trial and have signed information consent. Exclusion Criteria:Lymph node metastasis preoperatively.
* Tumors can not be resected .
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction, which may affect the treatment of Intrahepatic cholangiocarcinoma.
* Patients with a medical history of other malignant tumors.
* Subjects participating in other clinical trials.
* liver function:Child C.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | five years

SECONDARY OUTCOMES:
disease-free survival | five years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China